CLINICAL TRIAL: NCT03507296
Title: Spinal Kinematics Variability in Healthy Subjects and Patients With Chronic Low Back Pain in Different Functional Activities
Brief Title: Spinal Kinematics Variability
Status: Completed | Type: Observational
Sponsor: Haute Ecole de Santé Vaud (Other)
Responsible Party: Sponsor
Other Study IDs: VAR2017
Record Dates: First submitted 2018-03-14; First posted 2018-04-25 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic low back pain patients
- Asymptomatic subjects

SUMMARY:
This study will test the within and between day variability of spinal kinematics and trunk muscle activity in healthy subjects and chronic low back pain patients during various daily-life activities.

DETAILED DESCRIPTION:
This study will test the within and between day variability of spinal kinematics and trunk muscle activity in healthy subjects and chronic low back pain patients during various daily-life activities. Participants will come twice to the motion laboratory. During the first session, participants will first perform different functional activities (V1), such as sit-to-stand, gait, lifting tasks, stepping up. Their spinal kinematics will be measured with a camera-based system (VICON) using a multi-segment spinal model and trunk muscles activity will be recorded with surface electromyography. After a break, participants will have to perform all the functional activities a second time (V2). These two measures (V1 and V2) will be used to determine the within day variability of spinal kinematics. Finally, all participants will come one week later (V3) to repeat all the measurements to determine the between day variability.

ELIGIBILITY:
Inclusion Criteria:

* sufficient French level to understand the instructions for the tests, the information sheet, the consent form and the questionnaires
* All chronic low back pain patients should present with non-specific low back pain (pain from lower ribs to gluteal folds) for more than 3 months.

Exclusion Criteria:

* pregnancy
* body mass index (BMI) that is above 32
* patients should not have any sign of specific low back pain such as the presence of infection, rheumatological or neurological diseases, spinal fractures, any known important spinal deformities, previous back surgery that limits spinal mobility, tumours
* high level of pain at the time of experiment that prevents repeated movements (severity and irritability)
* other concomitant pain or condition that could compromise the evaluation of spinal kinematics.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic low back pain patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Spinal kinematics | Change between measure 1 and measure 2 (30 minutes later)
  Range of movement at the lower lumbar, upper lumbar, lower thoracic and upper thoracic joints
Trunk muscle activity | Change between measure 1 and measure 2 (30 minutes later)
  Surface electromyography of paraspinal, rectus abdominis and external obliques muscles
Spinal kinematics | Change between measure 1 and measure 3 (day 7)
  Range of movement at the lower lumbar, upper lumbar, lower thoracic and upper thoracic joints
Trunk muscle activity | Change between measure 1 and measure 3 (day 7)
  Surface electromyography of paraspinal, rectus abdominis and external obliques muscles

SECONDARY OUTCOMES:
Pain intensity | Measure 1 (Day 0), Measure 3 (Day 7)
  Pain intensity will be quantified by the 11-point Numeric Pain Rating Scale. The scale range from 0 (no pain at all) to 10 (worst pain).
Disability | Measure 1 (Day 0), Measure 3 (Day 7)
  Disability will be quantified by the Patient Specific Functional Scale. The scale assessed three relevant activities for the patient and scores each activity between 0 (impossible to realize the activity) to 10 (capable of doing the activity normally).
Disability (ODI) | Measure 1 (Day 0), Measure 3 (Day 7).
  Oswestry Disability Questionnaire. Score between 0 (no disability) and 100.
Kinesiophobia | Measure 1 (Day 0), Measure 3 (Day 7).
  Tampa Scale of Kinesiophobia. The total score is between 17 (no kinesiophobia) to 68 (high level of kinesiophobia).
Catastrophizing | Measure 1 (Day 0), Measure 3 (Day 7).
  Pain Catastrophizing Scale. Score between 0 and 52 (high levels of catastrophizing).
Back Pain Attitudes Questionnaire | Measure 1 (Day 0), Measure 3 (Day 7).
  Back Pain Attitudes Questionnaire. Score between 34 (positive attitudes) and 170 (negative attitudes)
Fear | Measure 1 (Day 0), Measure 2 (Day 0), Measure 3 (Day 7).
  Fear scale measured before each movement or activity. Score between 0 (no fear) and 10 (high levels of fear).
Pain expectation | Measure 1 (Day 0), Measure 2 (Day 0), Measure 3 (Day 7).
  Pain expectation scale before each movement or activity. Score between 0 (no pain expected) and 10 (high levels of pain expected).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lausanne Hospitals, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Christe G, Redhead L, Legrand T, Jolles BM, Favre J. Multi-segment analysis of spinal kinematics during sit-to-stand in patients with chronic low back pain. J Biomech. 2016 Jul 5;49(10):2060-2067. doi: 10.1016/j.jbiomech.2016.05.015. Epub 2016 May 20. PMID 27262182
- [Background] Christe G, Kade F, Jolles BM, Favre J. Chronic low back pain patients walk with locally altered spinal kinematics. J Biomech. 2017 Jul 26;60:211-218. doi: 10.1016/j.jbiomech.2017.06.042. Epub 2017 Jul 5. PMID 28716466